CLINICAL TRIAL: NCT02111265
Title: The Comparison of Efficacy and Safety of Target Controlled Infusion of Propofol or Etomidate at General Anesthesia in Geriatric Patients --A Randomized Controlled Trial.
Brief Title: THe Comparison of Target Controlled Infusion of Propofol or Etomidate at General Anesthesia in Geriatric Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Collaborators: Chinese Medical Association (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SAHXJTUA01
Record Dates: First submitted 2014-04-09; First posted 2014-04-11 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Adrenal Suppression; Hemodynamic Instability
MeSH Terms: interventions — Remifentanil; cisatracurium; Sufentanil; Monitoring, Physiologic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol (Experimental): Target controlled infusion propofol, the effect compartment concentration is 3-4μg/ ml for induction and maintenance of anesthesia.
  Interventions: Drug: Remifentanil; Drug: Cisatracurium; Drug: Sufentanil; Device: Bispectral index(BIS) monitor
- Etomidate (Experimental): Target controlled infusion etomidate, the effect compartment concentration is 0.5-1.0μg/ ml for induction and maintenance of anesthesia.
  Interventions: Drug: Remifentanil; Drug: Cisatracurium; Drug: Sufentanil; Device: Bispectral index(BIS) monitor

INTERVENTIONS:
Drug: Remifentanil — 1. Remifentanil 0.1-0.2μg/ ( kg•min) is continuously pumped at steady speed for analgesia for induction and maintenance of anesthesia.
  2. Remifentanil is stopped before skin closure
  Other Names: Ruijie
Drug: Cisatracurium — 1. Cisatracurium 0.15 mg/kg for induction and 0.12 mg/kg/h continuous infusion for maintenance of anesthesia.
  2. Cisatracurium is stopped before skin closure.
Drug: Sufentanil — Before skin closure, remifentanil is stopped and sufentanyl 0.1μg/kg is given by intravenous injection.
Device: Bispectral index(BIS) monitor — BiS is maintained at 40-60 during anesthesia.

SUMMARY:
Compare the efficacy and safety of closed-loop target controlled infusion of propofol or etomidate at general anesthesia in geriatric patients

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Scheduled for Endotracheal intubated and general anesthesia for general surgery patients.
3. Age 60-75 yrs.
4. American Society of Anesthesia (ASA) classification I-II.
5. Expected time of surgery is less than 3 hours. -

Exclusion Criteria:

1. Body mass index is more than 36kg/m2.
2. Systolic blood pressure≥180 mm Hg or <90 mm Hg，diastolic blood pressure≥110 mm Hg or < 60 mm Hg.
3. Serious cardiac,cerebral,liver,kidney,lung, endocrine disease or sepsis.
4. Long term used hormone or adrenal suppression.
5. Allergy to trial drug or other contraindication.
6. Difficult airway occurred before,or difficult airway possibly occurred and difficult to extubation.
7. Abuse of narcotic analgesia or suspected.
8. Neuromuscular diseases.
9. Mentally unstable or has a mental illness.
10. Malignant Hyperthermia.
11. Pregnant or breast-feeding women.
12. Attended other trial past 30 days. -

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-04; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Effect Compartment Concentration | From the beginning of induction to paitens'left of PACU, up to 4 hours
  The effect compartment concentration of etomidate or propofol are recorded at three time points,including time that patient's loss of eyelash reflex,after 30 minutes of loss of eyelash reflex and when the patient is awake （call then open their eyes).

SECONDARY OUTCOMES:
vital signs | From the beginning of induction to skin closure, up to 3 hours
  Systolic blood pressure, diastolic blood pressure, heart rate, respiration rate, pulse oxygen saturation recorded every 5 minutes during the operation.
The amount of drugs | From the beginning of induction to skin closure, up to 3 hours
  The amount of narcotics, sedation and muscle relaxation used in general anesthesia arr recorded when the operation is finished.
Adrenal function | From entering the operating room to 48 h after induction of anesthesia.
  1. 3 ml blood sample is collected at 5 time points including before induction,30 minutes,2 hours,24 hours, 48 hours after induction;
  2. to examine the concentration of Cortisol, Aldosterone and ACTH in serum:

CONTACTS AND LOCATIONS:
Overall Officials: He Jiaxuan, Principal Investigator — Department of Anesthesia, Second Affiliated Hospital of Xi'an Jiaotong University